CLINICAL TRIAL: NCT01495481
Title: Dexmedetomidine Versus Adenosine: Electrophysiologic Effects and Therapeutic Use for Terminating Supraventricular Tachycardia
Brief Title: Dexmedetomidine and Adenosine: Therapeutic Use for SVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Gaurav Arora, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO11070129; PRE-11-010 (Other Grant/Funding Number: Hospira, Inc)
Record Dates: First submitted 2011-12-15; First posted 2011-12-20 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Supraventricular Tachycardia
Keywords: Supraventricular Tachycardia; SVT; Reentrant Tachycardia; Dexmedetomidine; Adenosine
MeSH Terms: conditions — Tachycardia, Supraventricular | interventions — Dexmedetomidine; Adenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adenosine and Dexmedetomidine (Experimental): Patients will receive adenosine and then dexmedetomidine for the termination of SVT
  Interventions: Drug: Dexmedetomidine; Drug: Adenosine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 2 mcg/kg, Intravenous push
  Other Names: Precedex
Drug: Adenosine — Stepwise incremental approach of adenosine starting at 0.2 mg/kg (max 6 mg) followed by 0.3 mg/kg (max 12 mg) if initial dose was unsuccessful

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of dexmedetomidine in the acute termination of Supraventricular Tachycardia (SVT).

DETAILED DESCRIPTION:
In 2006 the investigator found that dexmedetomidine, an alpha-2 adrenergic agonist with primarily sedative properties, possesses additional anti-arrhythmic properties. So far the investigator has found that dexmedetomidine has the ability to prevent or terminate arrhythmias like atrial ectopic tachycardia (85% success) and junctional ectopic tachycardia (75% success). The most dramatic effect however was observed in the acute termination of reentrant SVT with a success rate of > 96%. More importantly we found that dexmedetomidine terminates SVT without causing any sinus pause or asystole (frequently seen with adenosine) and thus avoiding the feeling of "impending doom". In this study adenosine is being compared head to head with dexmedetomidine in a cross over study, for both safety and efficacy when given for the termination of SVT in the electrophysiology (EP) lab. Additional EP parameters will be measured to elucidate the exact site of dexmedetomidine's mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 5 - 30 years old, who are scheduled for cardiac electrophysiology study for evaluation of reentrant SVT

Exclusion Criteria:

* Severe Heart Failure
* Presence of of any other antiarrhythmic medication within 24 hours of enrollment
* Third degree heart block
* Sick Sinus Syndrome

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Arora, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Childrens Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chrysostomou C, Beerman L, Shiderly D, Berry D, Morell VO, Munoz R. Dexmedetomidine: a novel drug for the treatment of atrial and junctional tachyarrhythmias during the perioperative period for congenital cardiac surgery: a preliminary study. Anesth Analg. 2008 Nov;107(5):1514-22. doi: 10.1213/ane.0b013e318186499c. PMID 18931208
- [Background] Chrysostomou C, Sanchez-de-Toledo J, Wearden P, Jooste EH, Lichtenstein SE, Callahan PM, Suresh T, O'Malley E, Shiderly D, Haney J, Yoshida M, Orr R, Munoz R, Morell VO. Perioperative use of dexmedetomidine is associated with decreased incidence of ventricular and supraventricular tachyarrhythmias after congenital cardiac operations. Ann Thorac Surg. 2011 Sep;92(3):964-72; discussion 972. doi: 10.1016/j.athoracsur.2011.04.099. PMID 21871284

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 22 patients recruited received both adenosine and dexmedetomidine. Adenosine was administered first ,and then SVT was reinduced. Once SVT was reinduced, dexmedetomidine was administered.
  The washout period was not constant because it was dependent upon the reinduction of SVT, but it was generally less than 10 min.
Groups:
- Adenosine and Dexmedetomidine: Patients will receive adenosine for termination of SVT, and then dexmedetomidine for the termination of supraventricular tachycardia (SVT) and comparison will be made for efficacy and safety.
Period: Adenosine
Arm/Group | Adenosine and Dexmedetomidine
Started | 22 (Patients first received adenosine and then dexmedetomidine.)
Completed | 22
Not Completed | 0
Period: Washout
Arm/Group | Adenosine and Dexmedetomidine
Started | 22
Completed | 22
Not Completed | 0
Period: Dexmedetomidine
Arm/Group | Adenosine and Dexmedetomidine
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Adenosine and Dexmedetomidine: Patients will receive both adenosine and dexmedetomidine for the termination of SVT.
Arm/Group | Adenosine and Dexmedetomidine
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Termination of SVT
Description: Number of participants with SVT Termination within 3 minutes of medication administration
Time Frame: Within 3 minutes
Measure: Number; unit: participants
Groups:
- Dexmedetomidine: Patients will receive dexmedetomidine for the termination of SVT
  Dexmedetomidine: Dexmedetomidine 1 mcg/kg, Intravenous push
- Adenosine: Patients will receive Adenosine for the termination of SVT
  Adenosine: stepwise incremental approach of adenosine starting at 0.2 mg/kg (max 6 mg) followed by 0.3 mg/kg (max 12 mg) if initial dose was unsuccessful
Arm/Group | Dexmedetomidine | Adenosine
Number analyzed (Participants) | 22 | 22
participants | 16 | 21

2. Secondary Outcome: Number of Participants With Sinus Pause >2.5 Sec After Termination of SVT
Description: Evaluation of the number of participants with sinus pause > 2.5 sec, after dexmedetomidine vs. adenosine induced SVT termination
Time Frame: 1 minute
Measure: Number; unit: participants
Groups:
- Dexmedetomidine: Patients will receive dexmedetomidine for the termination of supraventricular tachycardia (SVT)
  Dexmedetomidine: Dexmedetomidine 2 mcg/kg, Intravenous push
Arm/Group | Dexmedetomidine | Adenosine
Number analyzed (Participants) | 22 | 22
participants | 0 | 16

3. Secondary Outcome: Number of Participants With Tachyarrhythmias After Medication Administration
Description: Number of participants with tachyarrhythmias, including Ventricular (Ventricular Tachycardia & Fibrillation)and supraventricular (Atrial Flutter & Fibrillation) after dexmedetomidine vs. adenosine administration
Time Frame: 10 minutes
Measure: Number; unit: participants
Groups:
- Dexmedetomidine: Patients will receive dexmedetomidine for the termination of supraventricular tachycardia (SVT)
  Dexmedetomidine: Dexmedetomidine 1 mcg/kg, Intravenous push
Arm/Group | Dexmedetomidine | Adenosine
Number analyzed (Participants) | 22 | 22
participants | 0 | 0

4. Secondary Outcome: Number of Participants With Hypotension by Non-invasive Cuff in First 10 Minutes After Medication Administration
Description: Blood pressure changes after dexmedetomidine vs. adenosine. Blood pressure measured by non-invasive cuff prior to medication administration, and then at 1 min, 3 min, 5 min after medication administration. Number of participants with a significant drop in blood pressure (mmHg) compared to baseline would be counted for hypotension.
Time Frame: 10 minutes
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine | Adenosine
Number analyzed (Participants) | 22 | 22
participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine | Adenosine
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No